CLINICAL TRIAL: NCT01547949
Title: Efficacy of Tart Cherry Juice in Reducing Muscle Injury and Biomarkers of Muscle Damage Among Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Cherry Research Committee (Other)
Responsible Party: Principal Investigator, Kerry Kuehl, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: e7220
Record Dates: First submitted 2012-02-24; First posted 2012-03-08 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Inflammation; Pain
Keywords: pain; inflammation; muscle damage
MeSH Terms: conditions — Inflammation; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tart cherry juice (Experimental)
  Interventions: Dietary Supplement: tart cultivar Montmorency cherry juice
- cherry flavored fruit drink (Placebo Comparator)
  Interventions: Dietary Supplement: placebo cherry fruit drink

INTERVENTIONS:
Dietary Supplement: tart cultivar Montmorency cherry juice
  Arms: tart cherry juice
Dietary Supplement: placebo cherry fruit drink
  Arms: cherry flavored fruit drink

SUMMARY:
The purpose of this study is to assess the effects of tart cherry juice to reduce serum biomarkers of inflammation and reduce muscle soreness in healthy adults who undergo a bout of controlled eccentric exercise.

DETAILED DESCRIPTION:
Numerous antioxidant and anti-inflammatory agents have been identified in tart cherries, and a study among healthy, non-exercising individuals demonstrated that tart cherries decreased post-exercise weakness and muscle pain. The purpose of this study is to assess the analgesic and myoprotective effects of tart cherry juice among healthy subjects in a randomized, placebo controlled, double-blind, crossover design trial. Fifteen healthy individuals will perform a bout of eccentric elbow flexion contractions (2 x 10 near maximum), and will then ingest 10 fl oz of a cherry juice or a placebo juice twice a day for four days, beginning immediately post exercise. Before and after exercise, and for three days following the eccentric exercise, blood will be drawn to measure serum biomarkers of muscle damage and muscle soreness will be recorded. The protocol will be repeated after a 9-10 day washout period with subjects consuming the alternative juice for the second trial. The opposite arm will perform the eccentric exercise for the second bout to avoid the repeated bout protective effect. The study's outcomes are 1) to assess changes in serum biomarkers of muscle damage, and 2) to assess changes in muscle soreness.

ELIGIBILITY:
Inclusion Criteria:

* no regular upper body strength training
* no elbow flexor pain, no history of elbow or shoulder injury
* ability and willingness not to take any anti-inflammatory or pain relieving drugs during the course of the study, not to seek any other treatment for any symptoms of muscle damage directly resulting from the exercises performed as part of the study, and not to exercise their upper extremities during the study.

Exclusion Criteria:

* individuals who have used or are using antiepileptic drugs for pain, acupuncture, or transcutaneous electrical nerve stimulation within 3 weeks before enrollment
* recent use (within 5 half-lives) of topical medications/anesthetics, muscle relaxants, tender point anesthetic injections within 2 months
* systemic steroid use within 3 months
* any investigational drug/device use in the prior 30 days
* individuals who have Type 1 or Type 2 Diabetes
* individuals who are pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Lactate | duration of intervention, average of 18 days per participant
  Primary outcomes include measurement of serum and plasma biomarkers that provide a generalized measurement of inflammatory activity; these include Creatine Kinase (CK), Aspartate aminotransferase (AST), Lactate dehydrogenase (LDH), and lactate.
Creatine Kinase | duration of intervention, average of 18 days per participant
  Primary outcomes include measurement of serum and plasma biomarkers that provide a generalized measurement of inflammatory activity; these include Creatine Kinase (CK), Aspartate aminotransferase (AST), Lactate dehydrogenase (LDH), and lactate.
Aspartate aminotransferase | duration of intervention, average of 18 days per participant
  Primary outcomes include measurement of serum and plasma biomarkers that provide a generalized measurement of inflammatory activity; these include Creatine Kinase (CK), Aspartate aminotransferase (AST), Lactate dehydrogenase (LDH), and lactate.
Lactate dehydrogenase | duration of intervention, average of 18 days per participant
  Primary outcomes include measurement of serum and plasma biomarkers that provide a generalized measurement of inflammatory activity; these include Creatine Kinase (CK), Aspartate aminotransferase (AST), Lactate dehydrogenase (LDH), and lactate.

SECONDARY OUTCOMES:
Secondary outcomes includes measurement of physical symptoms of exercise-induced muscle damage and soreness as measured by a muscle myometer. | duration of intervention, average of 18 days per participant

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Kuehl, MD, DrPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States